CLINICAL TRIAL: NCT00574522
Title: Phase 1 Study to Evaluate the Efficacy of Using Energy Specific Far Infrared Radiation Treatment for HIV/AIDS
Brief Title: Energy Specific Far Infrared Radiation Treatment for AIDS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Kwasi Donyina, Ph.D./Founder & President, Centre for Incurable Diseases, GAAD Medical Research Institute Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-HIV-CTP1
Record Dates: First submitted 2007-12-12; First posted 2007-12-17 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; Radiation; Far infrared; Treatment; Acquired Immunodeficiency Syndrome; Complimentary therapies
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Infrared Radiation, wavelength between 5 and 20 microns
  Interventions: Radiation: Far infrared

INTERVENTIONS:
Radiation: Far infrared — Far infrared radiation with the wavelength between 5μm and 20μm for 30 to 40 minutes per session.

SUMMARY:
The investigators are proposing that energy specific electromagnetic radiation of the central nervous system, the viscera and the endocrine system has the potential to enhance the immune system; thereby enhancing the production of killer cells to fight and destroy the human immunodeficiency virus.

DETAILED DESCRIPTION:
Acquired immune deficiency syndrome or acquired immunodeficiency syndrome (AIDS or Aids) is a collection of symptoms and infections resulting from the specific damage to the immune system caused by the human immunodeficiency virus (HIV) in humans. The late stage of the condition leaves individuals prone to opportunistic infections and tumors. Although treatments for AIDS and HIV exist to slow the virus' progression, there is no known cure.

The investigators are postulating that energy specific electromagnetic radiation of the central nervous system, the viscera and the endocrine system has the potential to enhance the immune system; thereby enhancing the production of CD4+ T cells and other killer cells to fight and destroy the human immunodeficiency virus.

The primary end point is to determine the therapeutic effects of far infrared radiation (5μm to 20μm wavelength) on HIV/AIDS.

ELIGIBILITY:
Inclusion Criteria:

* 1 Year and above

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
The primary end point is to determine the therapeutic effects of far infrared radiation (5μm to 15μm wavelength) on HIV/AIDS. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Principal Investigator — GAAD Medical Research Institute Inc.; Kwasi Donyina, Ph.D., Study Director — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada